CLINICAL TRIAL: NCT01674764
Title: Prognostic Factors and Therapeutic Effects of Surgical Treatment for Traumatic Spinal Column Injury With Spinal Cord Injury: A Prospective, Observational European Multi-center Study.
Brief Title: Surgical Treatment for Spinal Cord Injury
Acronym: SCI-POEM
Status: Completed | Type: Observational
Sponsor: AOSpine Europe (Industry)
Responsible Party: Sponsor
Other Study IDs: SCI-POEM
Record Dates: First submitted 2012-08-22; First posted 2012-08-29 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Acute Spinal Cord Injury of Traumatic Origin (tSCI)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Early surgical intervention = Cohort 1: ≤ 12 hours after the tSCI
  Interventions: Procedure: Early surgical intervention
- Late surgical intervention = Cohort 2: > 12 hours and < 14 days after the tSCI
  Interventions: Procedure: Late surgical intervention

INTERVENTIONS:
Procedure: Early surgical intervention — Open surgical stabilization and decompression (anterior, posterior or circumferential); and/or Closed reduction and external fixation
  Other Names: ≤ 12 hours after the tSCI
  Groups: Early surgical intervention = Cohort 1
Procedure: Late surgical intervention — Open surgical stabilization and decompression (anterior, posterior or circumferential); and/or Closed reduction and external fixation
  Other Names: > 12 hours and < 14 days after the tSCI
  Groups: Late surgical intervention = Cohort 2

SUMMARY:
Despite many years of research, an incomprehensible amount of scientific efforts worldwide and billions of dollars invested, no effective therapy resulting in major neurological or functional recovery is available to date for traumatic spinal cord injury (tSCI). Although there is increasing experimental evidence from animal models that surgical decompression of the spinal cord improves recovery after tSCI, clinical studies have not shown conclusive data yet. The main explanations for this lack of convincing evidence are relatively small sample sizes in previous studies, their predominantly retrospective nature, suboptimal measurement methods for the assessment of neurological deficits, and inappropriate recording and documentation of potential confounding factors.

DETAILED DESCRIPTION:
Although injuries to the spinal column represent a relatively small proportion of all traumatic injuries, spinal injuries have one of the highest impacts on functional outcomes and employment status. Even more than an injury of the spinal column, traumatic spinal cord injury (tSCI) is a devastating disorder severely affecting patients' physical and psychosocial well-being. The incidence of tSCI is estimated to be 11 to 53 new cases per million population per year.

This is a multi-center, prospective, observational cohort study to evaluate if early (≤ 12 hours after the tSCI) surgical decom¬pression is superior to late (> 12 hours and < 14 days after the tSCI) in improving neurologic motor outcomes in patients with acute traumatic spinal cord injury.

The study will enroll 300 patients with anticipated 1:2 ratio of early vs. late surgery. This CIP is not limited to cervical spinal cord injuries, does not consider a diagnostic MRI as mandatory and will be conducted in a European setting where patients are generally transported more swiftly to the treating institution when compared to other geographic regions in the world.

Patients will be evaluated according to the schedule set forth in this CIP. The schedule includes evaluations at pre-surgery, post-surgery, 72 hours post injury, 12 weeks ± 2 weeks; 6 months ± 30 days; 1 year ± 30 days. The enrollment period is expected to be approximately 36 months and subjects will be followed-up for 12 months for the evaluation of the primary endpoint. The study duration is approximately 48 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosis of blunt spinal column injury and spinal cord injury, including conus medullaris and/or cauda equina injuries
* Pre-surgery ASIA grade A, B, C or D
* Less than 14 days between the injury and surgery
* Ability to understand patient information / informed consent form
* Willingness and ability to participate in the clinical investigation and FU procedures (FUs)
* Informed consent according to local legislations and applicable guidelines

Exclusion Criteria:

* Traumatic brain injury: Glasgow Coma Scale (GCS) ≤ 13
* Diagnosis of subclinical or clinical polyneuropathy (eg. presence of bilateral impairment of strength, sensation, and/or deep tendon reflexes with symmetrical and distal distribution and/or neurophysiological abnormalities)
* Spinal cord injury caused by a penetrating injury
* Non-traumatic or pathologic fractures or cord compression (eg, tumor or infection)
* Unable to cooperate with physical examination (pre-operative, ≤ 2 weeks) because of cognitive impairment, as assessed by the examiner
* Previous spinal column or spinal cord injury
* Diagnosis of spondyloarthropathy (inflammatory or non-inflammatory)
* Morbid Obesity: Body Mass Index (BMI) > 35
* Any severe systemic disease that may have an influence on motor function (eg, polyneuropathy)
* ASA classification score ≥ 4
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment
* Pregnancy at the time of inclusion
* Prisoner
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll 300 patients with anticipated 1:2 ratio of early vs. late surgery. This CIP is not limited to cervical spinal cord injuries, does not consider a diagnostic MRI as mandatory and will be conducted in a European setting where patients are generally transported more swiftly to the treating institution when compared to other geographic regions in the world.
Sampling Method: Non-Probability Sample
Enrollment: 297 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in American Spinal Injury Association Lower Extremities Motor Score (ASIALEMS) between pre-surgery and 1-year post-surgery FU | Between pre-surgery and 1-year post-surgery

SECONDARY OUTCOMES:
Change in American Spinal Injury Association Motor Score (ASIAMS) between pre-surgery and 1-year FU | Pre-surgery and 1-year FU
Change in American Spinal Injury Association Upper Extremities Motor Score (ASIAUEMS) between pre-surgery and 1-year FU | Between pre-surgery and 1-year FU
Change in American Spinal Injury Association Impairment Scale (AIS) between pre-surgery and 1-year FU | Between pre-surgery and 1-year FU
Change in American Spinal Injury Association Sensory Score (ASIASS) between pre-surgery and 1-year FU | Between pre-surgery and 1-year FU
Spinal Cord Independency Measure (SCIM) at the 6-month and 1-year FU | 6-month and 1-year FU
Change in quality of life using the Short version of the World Health Organization Quality-of-Life questionnaire (WHOQOL-BREF) between pre-injury and 1-year FU | Pre-injury and 1-year FU
Rate of treatment related adverse events, as assessed by an independent evaluator | Until the 1-year FU

CONTACTS AND LOCATIONS:
Overall Officials: Allard JF Hosman, MD, PhD, Principal Investigator — Medical Co-Director Spine Unit, Radboud University Medical Centre, 6500 Nijmegen, The Netherlands
Locations (17):
- Medical University Innsbruck, Innsbruck, Austria
- National Institute of Emergency Medicine "N.I. Pirogov", Sofia, Bulgaria
- Teaching Hospital Sisiters of Charity, Zagreb, Croatia
- Hôspital P. Wertheimer, Lyon, France
- Germany (2):
  - BG Unfallklinik Frankfurt, Frankfurt
  - Berufsgenossenschaftliche Unfallklinik Ludwigshafen, Ludwigshafen
- Mater Misericordiae University Hospital, Dublin, Ireland
- Italy (2):
  - Ospedale Maggiore, Bologna
  - Policlinico Umberto Primo, Rome
- Netherlands (2):
  - University Medical Center St. Radboud, Nijmegen
  - University Medical Center Utrecht, Utrecht
- Spitalul "Sfanta Treime", Iași, Romania
- Clinical Center Vojvodina, Novi Sad, Serbia
- Gazi University Faculty of Medicine, Ankara, Turkey (Türkiye)
- United Kingdom (3):
  - King's College Hospital, London
  - Queens's Medical Centre Campus, Nottingham
  - Nuffield Orthopaedic Centre Headington, Oxford

REFERENCES:
- [Derived] Romijn P, Kussige PGP, van Hooff ML, Evaniew N, van de Meent H, van Middendorp JJ, Pouw MH, Hosman AJF. Early versus late surgical decompression in acute traumatic spinal cord injury: does it impact the quality of life? Spinal Cord. 2025 Dec 27. doi: 10.1038/s41393-025-01165-y. Online ahead of print. PMID 41455816